CLINICAL TRIAL: NCT05755802
Title: Ultrasound-guided Shoulder Block Versus Pericapsular Nerve Group Block (PENG) for Postoperative Analgesia in Arthroscopic Shoulder Surgery: a Randomized Controlled Trial
Brief Title: Shoulder Block Versus Pericapsular Nerve Group Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PENGB for shoulder surgery
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Surgery
Keywords: Pericapsular nerve group block

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation, perform the block, and administer bupivacaine solution
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (PENG block) (Active Comparator): Ultrasound-guided PENG block will be performed under strict aseptic precautions and patient's arm will be placed in external rotation and abducted at 45 degrees.
  Interventions: Procedure: PENG block
- Group B (Shoulder block) (Active Comparator): Ultrasound-guided shoulder block will be performed under strict aseptic precautions with patient in semi-recumbent position with the operating arm on the contra-lateral shoulder.and then, the patients will be positioned in a semi-recumbent position with the arm slightly flexed and adducted at the elbow for axillary nerve block.
  Interventions: Procedure: Shoulder block

INTERVENTIONS:
Procedure: PENG block — A linear ultrasound probe will be placed longitudinally between the coracoid and the humeral head. After defining the humeral head, the tendon of the subscapular muscle and the deltoid muscle over it, the needle will be inserted using the "in plane" technique. When the needle will have passed through the deltoid muscle and touched the subscapularis tendon, a bone-like hard tissue will be felt and the needle could not be advanced further. The needle tip will be placed between the deltoid muscle and subscapularis tendon, and the injectate will be slowly administered.
  Arms: Group A (PENG block)
Procedure: Shoulder block — The probe will be kept over the scapular spine to identify the trapezius and the supraspinatus muscle. Then, it Will be moved laterally to identify the concavity of the supraspinatus fossa and the hyper-echoic fascia of the supraspinatus muscle. In the concavity of the fossa, the suprascapular artery and the suprascapular nerve run in close proximity. A 50 mm nerve block needle will be used in the long axis view for the block. After confirming extravascular placement of the needle, injectate will be given below the supraspinatus fascia and then during axillary nerve block,The posterior surface of the humerus will be visualised in the short axis view. So, the circumflex artery will be visualised longitudinally. After confirming extra-vascular placement of the needle, injectate will be given into space.
  Arms: Group B (Shoulder block)

SUMMARY:
Effective analgesia in arthroscopic shoulder surgery is a major concern and is essential for all aspects of the patient's recovery. The aim of this study is to assess the quality of pain relief in patients who will undergo arthroscopic shoulder surgeries receiving either shoulder block versus PENG block comparing and evaluating the differences between the two techniques.It is hypothesized that PENG block will be comparable to shoulder block as a promising effective alternative for analgesia for arthroscopic shoulder surgeries with fewer side effects. It is suggested that the PENG block can be safely applied for analgesia.

DETAILED DESCRIPTION:
Effective analgesia in arthroscopic shoulder surgery is a major concern and is essential for all aspects of the patient's recovery. Multimodal pain management is recommended for early postoperative pain control. Regional anesthesia is preferred in shoulder surgery as an effective means of providing anesthesia and postoperative analgesia. Commonly used techniques for shoulder surgery include interscalene brachial plexus (ISB) blocks, continuous ISB (CISB) blocks, suprascapular nerve blocks (SSB), supraclavicular nerve blocks (SCB), local infiltration (LI), and ISB with adjuvants.Interscalene brachial plexus (ISB) block is considered the analgesic technique of choice for shoulder surgery. Shoulder block which is combination of suprascapular nerve block and axillary nerve block has been recently proposed as an alternative anesthetic and postoperative analgesic modality in this patient population. These two nerve blocks cause the loss of the sensory innervation of the shoulder. Shoulder block is advantageous to the interscalene brachial plexus block since it does not lead to respiratory dysfunction due to phrenic nerve palsy or other serious complications.The pericapsular nerve group (PENG) block may be safely applied for both partial anesthesia and analgesia in selected shoulder surgery cases. It did not cause motor block or pulmonary complications, nor result in muscle laxity, blocking only the shoulder and the upper third of the humerus. PENG block has been studied extensively in hip surgeries but its place in shoulder surgeries is not yet clear. Therefore, this study will be conducted to compare efficacy of ultrasound guided shoulder block with PENG block for postoperative analgesia in patients undergoing arthroscopic shoulder surgeries.

The aim of this study:

assess the quality of pain relief in patients who will undergo arthroscopic shoulder surgeries receiving either shoulder block versus PENG block comparing and evaluating the differences between the two techniques.

Sample Size Calculation:

Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 11.0.4 for windows (2011) with time to first analgesic request as the primary outcome. Using the results published by Pani et al 2019 with the mean time to first analgesic request in shoulder block group was (5.9 ± 1.2 hours) Using a two-sided two-sample unequal-variance t-test, sample size of 40 patients is needed to achieve 90% power to detect 20 % difference in time to first analgesic request. Using a two-sided hypothesis test with a significance level of 0.05. A 10% drop out is considered, so a total of 46 patients will be enrolled (23 in each group) in this study.

Methods:

The study will be conducted in Mansoura university hospital on Forty six patients who will be scheduled for arthroscopic shoulder surgery under general anesthesia. They will be randomly assigned to two equal groups (PENG group and shoulder block group) according to computer-generated table of random numbers using the permuted block randomization method. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent. A written informed consent will be obtained from all study subjects after ensuring confidentiality. The study protocol will be explained to all patients after enrollment into the study along with VAS after enrollment into the study. Basic demographic characters including age, sex, and weight will be recorded. In both groups, The PENG and shoulder block procedures will be performed in the preoperative regional room under strict aseptic conditions using 30 ml 0.25% bupivacaine.

Statistical Methods:

The collected data will be coded, processed, and analyzed using SPSS(Statistical Package for the Social Sciences) program (version 22) for Windows. Normality of numerical data distribution will be tested by Shapiro-Wilk test. Continuous data of normal distribution will be presented as mean ± SD(standard deviation) and compared with the unpaired student's t test. Non-normally distributed data will be presented as median (range) and compared with the Mann-Whitney U test. Repeated measures ANOVA will be used for comparisons within the same group. Categorical data will be presented as number (percentage) and compared with the Chi-square test. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) 1 or 2 patients.
* Scheduled for elective unilateral shoulder arthroscopy.

Exclusion Criteria:

* Patient's refusal.
* Altered mental status or un-cooperative patients.
* History of known sensitivity to the used anesthetics.
* Bleeding or coagulation diathesis.
* Infection or redness at the injection site.
* Significant cardiac dysfunction, hepatic, or renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
First analgesic request | Up to 24 hours after the procedure
  The time of the first analgesic request for fentanyl will be recorded.

SECONDARY OUTCOMES:
Visual analogue score (VAS) for pain assessment | Up to 24 hours after the procedure
  VAS score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) will be assessed every two hours for 24 hours after the procedure.
Total analgesic requirements of fentanyl | Up to 24 hours after the procedure
  The amount of fentanyl consumption given as a rescue analgesia to patients will be measured all over the 24 hours.
Heart rate (HR) | During the procedure
  HR will be recorded every 30min till the end of the procedure.
Mean arterial blood pressure (MAP) | During the procedure
  MAP will be recorded every 30min till the end of the procedure.
Adverse effects | Up to 24 hours after the procedure
  Pneumothorax, respiratory depression, nausea, vomiting, hematoma, or allergic reactions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amany H EL-Deeb, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Casas Reza P, Dieguez Garcia P, Gestal Vazquez M, Sampayo Rodriguez L, Lopez Alvarez S. Pericapsular nerve group block for hip surgery. Minerva Anestesiol. 2020 Apr;86(4):463-465. doi: 10.23736/S0375-9393.20.14166-X. Epub 2020 Jan 28. No abstract available. PMID 32000476
- [Result] van Erp JHJ, Ostendorf M, Lansdaal JR. Shoulder surgery in beach chair position causing perioperative stroke: Four cases and a review of the literature. J Orthop. 2019 May 27;16(6):493-495. doi: 10.1016/j.jor.2019.05.009. eCollection 2019 Nov-Dec. PMID 31680738
- [Result] Kapukaya F, Ekinci M, Ciftci B, Atalay YO, Golboyu BE, Kuyucu E, Demiraran Y. Erector spinae plane block vs interscalene brachial plexus block for postoperative analgesia management in patients who underwent shoulder arthroscopy. BMC Anesthesiol. 2022 May 12;22(1):142. doi: 10.1186/s12871-022-01687-5. PMID 35550031
- [Result] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Result] Pani N, Routray SS, Pani S, Mallik S, Pattnaik S, Pradhan A. Post-operative analgesia for shoulder arthroscopic surgeries: A comparison between inter-scalene block and shoulder block. Indian J Anaesth. 2019 May;63(5):382-387. doi: 10.4103/ija.IJA_65_19. PMID 31142882
- [Result] Patel MS, Abboud JA, Sethi PM. Perioperative pain management for shoulder surgery: evolving techniques. J Shoulder Elbow Surg. 2020 Nov;29(11):e416-e433. doi: 10.1016/j.jse.2020.04.049. Epub 2020 Jun 9. PMID 32844751
- [Result] Sahin A, Baran O, Cetin MU, Gultekin A, Arar MC. Combined suprascapular nerve block and axillary nerve block approach vs. peri-articular infiltration analgesia for postoperative pain management following arthroscopic shoulder surgery: a randomized clinical trial. Eur Rev Med Pharmacol Sci. 2022 Dec;26(24):9117-9125. doi: 10.26355/eurrev_202212_30661. PMID 36591824
- [Result] Sripada R, Bowens C Jr. Regional anesthesia procedures for shoulder and upper arm surgery upper extremity update--2005 to present. Int Anesthesiol Clin. 2012 Winter;50(1):26-46. doi: 10.1097/AIA.0b013e31821a0284. PMID 22227421